CLINICAL TRIAL: NCT02690948
Title: A Phase 1b Open Label Study of Pembrolizumab for Unresectable or Metastatic Basal Cell Carcinoma
Brief Title: Pembrolizumab With or Without Vismodegib in Treating Metastatic or Unresectable Basal Cell Skin Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anne Chang (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Anne Chang, Associate Professor of Dermatology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-34925; NCI-2015-01869 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 350 (Other: NCI); P30CA124435 (NIH); SKIN0031 (Other: OnCore)
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Skin Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — pembrolizumab; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab Monotherapy (Experimental): Participants who previously received vismodegib and subsequently progressed will receive pembrolizumab IV over 30 minutes on day 1. Cycles are every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab
- Pembrolizumab plus Vismodegib Combination Therapy (Experimental): Participants who have not progressed while receiving vismodegib will receive pembrolizumab IV over 30 minutes on day 1 and take vismodegib 150 mg by mouth daily. Cycles repeat every 21 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Vismodegib

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449
  Arms: Pembrolizumab plus Vismodegib Combination Therapy

SUMMARY:
This phase 1-2 trial studies how well pembrolizumab with or without vismodegib works in treating patients with skin basal cell cancer that has spread to other places in the body or cannot be removed by surgery. Monoclonal antibodies, such as pembrolizumab, are checkpoint inhibitors that stimulate immune response. Vismodegib may stop the growth of tumor cells by blocking signals needed for cell growth.

DETAILED DESCRIPTION:
This study is a non-randomized evaluation of pembrolizumab as a treatment for unresectable or metastatic basal cell carcinoma (BCC). Participants are assigned to treatment with pembrolizumab plus vismodegib or pembrolizumab monotherapy on the basis of suitability for treatment with smoothened (SMO) inhibitors such as vismodegib. Prospective participants who have progressed on vismodegib, are intolerant to or have a medical contra-indication to vismodegib may receive pembrolizumab monotherapy. Because treatment is non-randomized, no comparison between treatment groups is conducted.

PRIMARY OBJECTIVE To assess the overall response rate (ORR) of unresectable or metastatic BCC patients to pembrolizumab with or without vismodegib (all evaluable patients) at 18 weeks

SECONDARY OBJECTIVES

* To assess the ORR of unresectable or metastatic BCC patients to pembrolizumab monotherapy at 18 weeks
* To assess the ORR of unresectable or metastatic BCC patients to pembrolizumab monotherapy at 9 weeks
* To assess ORR of unresectable or metastatic BCC patients to pembrolizumab plus vismodegib at 18 weeks
* To assess ORR of unresectable or metastatic BCC patients to pembrolizumab plus vismodegib at 9 weeks
* To assess the safety and tolerability of pembrolizumab (either monotherapy or combination therapy) for unresectable or metastatic BCC.
* To assess the duration of response after pembrolizumab (either monotherapy or combination therapy)
* Incidence and severity of adverse events
* Correlative studies including programmed death-ligand 1 (PD-L1) expression pre-treatment, lymphocytic infiltrates pre- and post-treatment, mutational analysis pre- and post-treatment

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically-proven basal cell carcinoma (BCC) in which curative resection is unlikely without significant morbidity, or have nodal or distantly metastatic disease which has progressed on vismodegib (Arm 1) or has achieved partial response or stable disease on smoothened inhibitor (Arm 2). Individuals who are intolerant or have a medical contra-indication to smoothened inhibitor will be enrolled into Arm 1.
* Have measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1
* ≥ 18 years of age on day of consent.
* Willing to provide tissue from a core or excisional biopsy of a tumor lesion up to 6 weeks (42 days) prior to initiation of treatment on Day 1, or availability of adequate archival specimens.
* Eastern Cooperative Oncology Group (ECOG) Performance Status = 0 or 1
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL, or ≥ 5.6 mmol/L, without transfusion or EPO dependency (within 7 days of assessment)
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance ≥ 60 mL/min for subject(s) with creatinine levels > 1.5 x ULN
* Serum total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN, OR ≤ 5 x ULN for subjects with liver metastases
* alanine aminotransferase (ALT) ≤ 2.5 x ULN, OR ≤ 5 x ULN for subjects with liver metastases
* Albumin ≥ 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy, in which case PT/INR must be within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy, in which case PTT must be within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or be willing to abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* If female, is postmenopausal; is surgically sterile; or agrees to use 2 acceptable methods of birth control throughout the trial, until 120 days after the last dose of treatment
* If female, agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Male with female partner of childbearing potential agrees to use adequate method of contraception throughout study, until 120 days after last dose of treatment or last blood draw.
* Willing and able to provide written informed consent/assent for the trial. Consent may be obtained by legally-authorized representative (LAR).

EXCLUSION CRITERIA

* Currently receiving investigational study therapy, or has received investigational study therapy, or used an investigational device, within 4 weeks of the first dose of treatment.
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (EXCEPTIONS: topical, intraarticular, intralesional, and inhaled steroids)
* Known history of active Bacillus Tuberculosis (TB) infection
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has received an anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1, or who has not recovered (ie, ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has received chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1, or who has not recovered (ie, ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. (EXCEPTION: Subjects with ≤ Grade 2 neuropathy may qualify for the study).
* If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Known additional malignancy that is progressing or requires active treatment. (EXCEPTIONS: basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer)
* Carcinomatous meningitis without consideration of clinical stability
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Intraarticular, inhaled, and intralesional doses of steroids are allowed at screening and during the study.
* Known history of, or any evidence of active, non-infectious pneumonitis that required steroids or current pneumonitis.
* Active infection requiring systemic therapy.
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding
* Expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1-2 antibodies).
* Has known active Hepatitis B (eg, HBsAg reactive) or Hepatitis C (eg, HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (eg, Flu-Mist) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lynn S Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.7 (11.2) | 61.9 (7.51) | 65.1 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The overall response rate (ORR) of participants with unresectable or metastatic basal cell carcinoma (BCC) after treatment with A) pembrolizumab monotherapy and B) pembrolizumab in combination with vismodegib, will be assessed as the percentage of participants with partial response (PR) or complete response (CR) as determined by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria, after 9 and 18 weeks of treatment. ORR is calculated as the ratio of patients with CR or PR as a percentage of the participants evaluable for OR.
  RECIST criteria:
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: 18 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy
Number analyzed (Participants) | 9 | 7
Percentage of participants | 44 [14 to 79] | 29 [4 to 71]

2. Secondary Outcome: Percentage of Participants Experiencing Adverse Events
Description: Incidence of Adverse Events is assessed as the percentage of participants receiving treatment who experience adverse events of any grade, in participants receiving A) pembrolizumab monotherapy and B) pembrolizumab in combination with vismodegib. Enrolled participants receiving at least one dose of study agent and with at least one follow-up evaluation will be included.
Time Frame: up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy
Number analyzed (Participants) | 9 | 7
percentage of participants | 100 | 100

3. Secondary Outcome: Related Adverse Events
Description: Adverse events were assessed for relationship to pembrolizumab treatment. The outcome is reported as the number (without dispersion) of Grade 3 or higher adverse events considered possibly, probably, or definitely-related to pembrolizumab treatment,.
Time Frame: up to 2 years
Measure: Number; unit: Related adverse events
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy
Number analyzed (Participants) | 9 | 7
Related adverse events | 1 | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: The duration of response (DOR) as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria in participants receiving A) pembrolizumab monotherapy and B) pembrolizumab in combination with vismodegib, assessed as the median value for subjects who complete 9 and 18 weeks of treatment.
  RECIST criteria:
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: up to 2 years
Measure: Median (Full Range); unit: Weeks
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy
Number analyzed (Participants) | 4 | 2
Weeks | 67.57 [31.43 to 82] | 52.78 [28 to 77.57]

5. Secondary Outcome: Overall Survival (OS)
Description: The overall survival (OS) participants with unresectable or metastatic basal cell carcinoma (BCC) after treatment with A) pembrolizumab monotherapy and B) pembrolizumab in combination with vismodegib, will be reported as the number and percentage of participants remaining alive 1 year after the start of treatment.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy
Number analyzed (Participants) | 9 | 7
Participants | 9 | 7

6. Secondary Outcome: Progression-free Survival (PFS)
Description: The progression-free survival (PFS) will be participants with unresectable or metastatic basal cell carcinoma (BCC) after treatment with A) pembrolizumab monotherapy and B) pembrolizumab in combination with vismodegib, will be reported as the percentage of participants without progression 1 year after the start of treatment.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy
Number analyzed (Participants) | 9 | 7
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Pembrolizumab Monotherapy | Pembrolizumab Plus Vismodegib Combination Therapy
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/9 | 2/7
Other Adverse Events (participants affected / at risk) | 9/9 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Monotherapy (N=9) | Pembrolizumab Plus Vismodegib Combination Therapy (N=7)
Hypertension (Vascular disorders) | 1 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, right shoulder four quarter amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures - tumor resection (Surgical and medical procedures) | 0 (0) | 1 (1)
Infections and infestations - Other, Peri-incisional cellulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab Monotherapy (N=9) | Pembrolizumab Plus Vismodegib Combination Therapy (N=7)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 6 (6) | 3 (3)
Fever (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (6) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder -Other, muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder -Other, gout (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Eye disorders - Other, ptosis (Eye disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, seborrheic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Verruca (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, psoraisis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Eye Erosion (Eye disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 2 (3) | 1 (1)
Cardiac disorders - Other, Premature ventricular contraction (Cardiac disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood and lymphatic system disorders-Other, Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Infections and infestations -Other, Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (1) | 1 (2)
Surgical and medical procedures - Other, Elective Surgery-Foot (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Root Canal (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Mohs Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, Skin tag removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Other, Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) -Other, squamous cell carcinoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT02690948/Prot_SAP_000.pdf